CLINICAL TRIAL: NCT03487692
Title: Diabetes MESSAGES (Medical Care, Education, Social Support, And Goal-setting to Empower Self-management): Implementing Diabetes Group Visits and Text Messaging in Community Health Centers
Brief Title: Medical Care, Education, Social Support, And Goal-setting to Empower Self-management for Diabetes
Acronym: MESSAGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Midwest Clinicians' Network (Unknown); CareMessage (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB17-1385
Record Dates: First submitted 2018-03-21; First posted 2018-04-04 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; group visit; shared medical appointment; text messaging
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2018 Training Cohort (Experimental): 10 health centers will be randomized to the 2018 Training Cohort. Teams from these health centers will be trained and will implement a 6 month diabetes group visit and text messaging intervention (Diabetes MESSAGES Program).
  Interventions: Other: Diabetes MESSAGES Program
- 2020 Training Cohort (Other): 10 health centers will be randomized to the 2020 Training Cohort. Prior to beginning training, these health centers will collect data on randomly selected patients receiving usual care to serve as the control group. After this first parallel group trial period, teams from these health centers will be trained and will implement the 6 month diabetes group visit and text messaging intervention during a second single group trial period (Diabetes MESSAGES Program (second trial)).
  Interventions: Other: Diabetes MESSAGES Program (second trial)

INTERVENTIONS:
Other: Diabetes MESSAGES Program — Health centers in the 2018 Training Cohort will enroll groups of 10-15 patients to attend 6 monthly diabetes group visits consisting of group education, social support, goal setting, and an individual medical visit for each patient. At the same time, patients will be enrolled in a 6-month interactive diabetes text messaging program. Patients will receive quarterly booster sessions for 1-2 years after the 6-month intervention period.
  Arms: 2018 Training Cohort
Other: Diabetes MESSAGES Program (second trial) — During the first trial period, health centers in the 2020 Training Cohort will collect data on patients receiving usual care. After the first trial period, health centers in the 2020 Training Cohort will enroll groups of 10-15 patients to attend 6 monthly diabetes group visits consisting of group education, social support, goal setting, and an individual medical visit for each patient. At the same time, patients will be enrolled in a 6-month interactive diabetes text messaging program. Patients will receive quarterly booster sessions for 1-2 years after the 6-month intervention period.
  Arms: 2020 Training Cohort

SUMMARY:
Diabetes group visits, shared appointments where patients receive self-management education in a group setting and have a medical visit, are a promising way to deliver high quality diabetes care. Group visits can improve glycemic control and decrease healthcare utilization. To date, no studies have systematically implemented a diabetes group visit intervention in a network of U.S. community health centers. The University of Chicago is partnering with Midwest Clinicians' Network (MWCN), a member organization of 130 health centers across ten Midwestern states. Approximately half of all Federally Qualified Health Centers in this region are affiliated with MWCN. The objectives of the study are [1] providers and staff at 20 health centers will have the requisite knowledge, skills, and motivation to implement a diabetes group visit plus text messaging intervention at their sites; [2] changes in diabetes processes of care; knowledge, attitudes, and skills for diabetes self-management; clinical outcomes; and health care utilization for patients participating in the diabetes group visit program will be evaluated; and [3] the diabetes group visit program will be available for dissemination among and use by health centers and healthcare providers at the local, state, regional, and national levels.

DETAILED DESCRIPTION:
UChicago and MWCN will recruit and enroll 20 health centers (HCs) to participate in a training intervention and to implement diabetes group visit and text messaging programs at their clinic sites. Each HC will assemble a team of 3-4 providers and staff to participate in the training. HCs will be randomized to one of two training cohorts. HC providers and staff will attend two in-person Learning Sessions in Chicago and a series of monthly webinars, recruit and enroll patients, implement a 6-month diabetes group visit and text messaging program plus subsequent booster sessions, complete periodic surveys and interviews, assist with data collection through patient surveys and chart abstraction, and present their program to peer HCs during Learning Sessions and to local stakeholders, state primary care organizations, or other professional groups. Each HC will enroll 15 patients in the group visit and text messaging program; the 2018 Training Cohort will do so immediately following their enrollment in the study and the 2020 Training Cohort will do so after 18 months. During the first 18 months, the 2020 Training Cohort will collect data from electronic health records (EHR) of randomly selected patients to serve as a control group. Changes in self-reported outcomes, diabetes processes of care, and clinical outcomes will be assessed for intervention patients from baseline through 2 year follow up, and processes of care and clinical outcomes will be compared for intervention vs. control participants. Capacity of HC providers and staff to conduct a group visit and text messaging intervention for patients with diabetes, as well as their confidence in identifying and addressing health disparities, will be evaluated through surveys and in-depth interviews. This study will expand knowledge of the barriers, facilitators, and perceived benefits and drawbacks of group visit and text messaging interventions and inform the development of a toolkit that will be disseminated to other HCs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* diagnosis of type 2 diabetes
* attended at least two appointments at the HC within the past year, with at least one of them being during the past six months
* last documented A1c result greater than or equal to 8.0% (test must have been done during the last 6 months)
* own a cellular phone with text messaging capabilities
* have the ability to read and send text messages
* English or Spanish speaking

Exclusion Criteria:

* pregnant or planning to become pregnant
* uncontrolled psychiatric problem
* dementia or other cognitive impairment
* hearing difficulties or severe physical disability that would prevent them from participation in group visit
* planning to relocate in the next year or leave the area during the group visit period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | change from baseline to 12 months

SECONDARY OUTCOMES:
Hemoglobin A1C | baseline, 6 month, and 18 month for intervention vs. control patients; 30 month for intervention patients only
Blood pressure | baseline, 6 month, and 18 month for intervention vs. control patients; 30 month for intervention patients only
Weight | baseline, 6 month, and 18 month for intervention vs. control patients; 30 month for intervention patients only
Cholesterol | baseline, 6 month, and 18 month for intervention vs. control patients; 30 month for intervention patients only
Diabetes processes of care | baseline, 6 month, and 18 month for intervention vs. control patients; 30 month for intervention patients only
  Receipt of recommended screenings, exams, referrals, and vaccinations
Medication management of diabetes | baseline, 6 month, and 18 month for intervention vs. control patients; 30 month for intervention patients only
  changes in prescribed diabetes medications for patients with inadequate diabetes control
Number of hypoglycemic events | baseline, 6 month, and 12 month for intervention patients only
Number of hospital admissions | baseline, 6 month, and 18 month for intervention vs. control patients; 30 month for intervention patients only
Number of primary care, specialist, and ER visits | baseline, 6 month, and 18 month for intervention vs. control patients; 30 month for intervention patients only
Smoking status | baseline, 6 month, and 12 month for intervention patients only
Health related quality of life (SF-12) | baseline, 6 month, and 12 month for intervention patients only
Depression (PHQ-2) | baseline, 6 month, and 12 month for intervention patients only
Summary of Diabetes Self-Care Activities Measure | baseline, 6 month, and 12 month for intervention patients only
Understanding of Diabetes Self-Management (Diabetes Care Profile) | baseline, 6 month, and 12 month for intervention patients only
Attitudes Towards Diabetes (Diabetes Care Profile) | baseline, 6 month, and 12 month for intervention patients only
Diabetes Distress Scale (DDS-2) | baseline, 6 month, and 12 month for intervention patients only
Diabetes Quality of Life Scale | baseline, 6 month, and 12 month for intervention patients only
Diabetes Self-Empowerment Scale | baseline, 6 month, and 12 month for intervention patients only
Diabetes Social Support Scale | baseline, 6 month, and 12 month for intervention patients only
Patient satisfaction with intervention | 6 month and 12 month for intervention patients only
CAHPS Overall Rating | baseline, 6 month, and 12 month for intervention patients only
  Patient satisfaction with overall care at health center
CAHPS Cultural Competency | baseline, 6 month, and 12 month for intervention patients only
  Patient satisfaction with cultural competency of care at health center
CAHPS Provider Communication | baseline, 6 month, and 12 month for intervention patients only
  Patient satisfaction with provider communication at health center

OTHER OUTCOMES:
Patient engagement | through study completion, an average of 2 years
  Attendance/participation in group visits, text messaging, and booster sessions
Health center provider/staff preparedness | change from pre- to post-training (from baseline to 1 month, 7 month, and 16 month)
  Capacity, confidence, motivation, perceived benefits and barriers
Health center provider/staff satisfaction | post-training (16 month)
  Satisfaction with training, group visits, and text messaging

CONTACTS AND LOCATIONS:
Overall Officials: Arshiya Baig, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No